CLINICAL TRIAL: NCT02447640
Title: An Open Label PET Imaging Study to Evaluate the mGlu5 Receptor Occupancy Following ADX48621 (Dipraglurant) Administration
Brief Title: PET Imaging Study to Evaluate the mGlu5r Occupancy Following ADX48621 (Dipraglurant) Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Addex Pharma S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ADX48621-104
Record Dates: First submitted 2015-04-02; First posted 2015-05-19 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: Volunteers
MeSH Terms: interventions — 6-fluoro-2-(4-(pyridin-2-yl)but-3-yn-1-yl)imidazo(1,2-a)pyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Experimental): A receptor occupancy dose curve will be obtained by using an adaptive design in this arm.
  Interventions: Drug: ADX48621; Radiation: [18F]FPEB
- Part 2 (Experimental): In this arm, the time course of the receptor occupancy will be studied for the dose which gives 70% receptor occupancy as determined in Part 1.
  Interventions: Drug: ADX48621; Radiation: [18F]FPEB

INTERVENTIONS:
Drug: ADX48621 — ADX4862, an investigational compound, is a potent, selective, negative allosteric modulator of the metabotropic glutamate receptor 5 (mGlu5 NAM).
  Other Names: dipraglurant
Radiation: [18F]FPEB — radiotracer used for PET scanning

SUMMARY:
This is an open label study, non-randomized, positron emission tomography (PET)study investigating mGlu5 receptor occupancy after single or two oral dosing of ADX48621 in healthy subjects using [18F]-FPEB as the radiotracer.

DETAILED DESCRIPTION:
This is an open label study, non-randomized, positron emission tomography (PET) study investigating mGlu5 receptor occupancy after single or two oral dosing of ADX48621 in healthy subjects using [18F]-FPEB . The study consists of 2 parts.

Part 1: A receptor occupancy dose curve will be obtained by using an adaptive design. Subjects will undergo two [18F]-FPEB PET imaging sessions: a baseline plus a scan after treatment with one dose of ADX48621. The second scan will be taken at Tmax for ADX48621 (1 hour post dose). 100 mg will be the initial dose as this has been proven to be efficacious in a P2A study in Parkinson's patients. This is an open label study, non-randomized, positron emission tomography (PET)study investigating mGlu5 receptor occupancy after single or two oral dosing of ADX48621 in healthy subjects using [18F]-FPEB as the radiotracer.The maximum dose to be given will be 200 mg.

Part 2: The time course of the receptor occupancy will be studied for the dose which gives 70% receptor occupancy as determined in Part 1. Two subjects will receive 2 doses of ADX48621 on 2 separate days and undergo three [18F]-FPEB PET imaging sessions: a baseline scan, post dose scan 1 and post dose scan 2. Subjects will be given ADX48621 one hour prior post dose scan 1. The 2nd dose will be given in the morning approximately 4-6 hours prior of the post dose scan 2. The post dose scan 2 will be performed in the afternoon. The maximum dose to be given will be 400 mg.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, 18-60 years old
* BMI of 18-32 kg/m2
* Female subjects must meet one of the following criteria:Surgically sterile (e.g. hysterectomy, or bilateral oophorectomy, tubal ligation) for at least 6 months prior to screening or Postmenopausal (no menstrual bleeding for at least 1 year prior to screening and confirmed by a plasma FSH level of > 40 IU/L) or Non-pregnant, non- lactating women of child-bearing potential and practicing contraception (e.g. hormonal birth control, intra uterine device, condom and spermicide)
* Able to comprehend and willing to sign an Informed Consent Form (ICF).

Exclusion Criteria:

* Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or any psychiatric disorder (as determined by the Investigator).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator.
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (except that appendectomy and hernia repair will be allowed).
* Use of any tobacco-containing or nicotine-containing products (including, but not limited to, cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to consent.
* Poor peripheral venous access.
* Participation in any clinical drug study within 30 days prior to dosing.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the maximum receptor occupancy and EC 50 for the receptor occupancy/ADX48621 plasma concentration relationship | During Day 1 PET scan
  This is composite

CONTACTS AND LOCATIONS:
Overall Officials: Dean F Wong, MD,PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States